CLINICAL TRIAL: NCT06407505
Title: The Effect of LI4 Acupressure on Perineal Pain and Postpartum Comfort During Episiotomy Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Derya Deniz, lecturer, Uskudar University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Labor Pain; Perineal Pain; Postpartum Comfort
Keywords: Acupressure, LI4 acupoint, Perineal pain, Postpartum comfort
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Our study was designed as a randomized, controlled, single-blind, placebo-designed experimental study.
Who Masked: Participant
Masking Description: The process will not know the group to which the patient belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure group (Experimental): During the episiotomy repair, the LI4 acupuncture point on the right hand of the participants in the experimental group will be compressed 10 times for 30 s in succession, followed by a 10 s break.
  Interventions: Other: Acupressure group
- Placebo Group (Placebo Comparator): A different point 1-1.5 cm away from the LI4 acupuncture point on the right hand of the participants in the placebo group will be compressed.
  Interventions: Other: Placebo group
- Control Group (No Intervention): Group receiving routine care.

INTERVENTIONS:
Other: Acupressure group — LI4 acupressure applied group.
  Other Names: LI4 acupressure group; experimental
  Arms: Acupressure group
Other: Placebo group — Group where acupressure was applied to an area 1.5 cm away at the LI4 acupressure point
  Arms: Placebo Group

SUMMARY:
The study was planned to evaluate the effect of LI4 acupressure application on perineal pain and postpartum comfort during episiotomy repair. Our study was designed as a randomized, controlled, single-blind and placebo design experimental study. The study is planned to be conducted in the maternity ward of Istanbul SBU Kanuni Sultan Süleyman Training and Research Hospital between May 1, 2024 and October 20, 2025. The sample of the study will consist of a total of 90 pregnant women who were hospitalized in the maternity ward and agreed to participate in the study. During the episiotomy repair, the LI4 acupuncture point on the right hand of the participants in the experimental group will be compressed 10 times for 30 seconds in succession and a 10-second break will be taken. A different point 1-1.5 cm away from the LI4 acupuncture point on the right hand of the participants in the placebo group will be pressed. No intervention will be applied to the control group.

DETAILED DESCRIPTION:
Background: Pain relief in the intrapartum period is important for maternal-fetal health. Studies in the literature have generally focused on the first stage of labor. When the labor process is considered as a whole, women may also experience pain during episiotomy repair. In recent years, traditional methods have become more preferred due to the side effects of pharmacologic treatments to relieve pain symptoms. Acupressure, one of the traditional methods, is used to relieve pain and various symptoms by applying pressure on acupuncture points with manual techniques. In the literature, LI4 acupressure is applied to relieve pain symptoms caused by various reasons. However, among the studies reviewed, no study was found to investigate the effect of LI4 acupressure application on perineal pain perceived during episiotomy repair and postpartum comfort level.

Objective: The study was planned to evaluate the effect of LI4 acupressure on perineal pain and postpartum comfort during episiotomy repair.

Materials and Methods: Our study was designed as a randomized, controlled, single-blind, placebo-designed experimental study. The study will be conducted in the maternity ward of Istanbul SBÜ Kanuni Sultan Süleyman Training and Research Hospital between May 1, 2024 and October 20, 2025. The sample of the study will consist of a total of 90 pregnant women (experimental group= 30, control group= 30, placebo group= 30) who were hospitalized in the maternity ward and agreed to participate in the study. During the episiotomy repair, the LI4 acupuncture point on the right hand of the participants in the experimental group will be compressed 10 times for 30 s in succession, followed by a 10 s break. The procedure will start with the first suturing. Vital signs will be taken just before the first suturing and after the suturing is completed. A different point 1-1.5 cm away from the LI4 acupuncture point on the right hand of the participants in the placebo group will be compressed. No intervention will be applied to the control group. Data will be obtained using the Pregnancy Identification Form, Visual Comparison Scale, Postpartum Comfort Scale, Labor Monitoring Form and McGill Pain Scale Short Form. The data obtained from the study will be analyzed in SPSS 23 statistical program in computer environment. In the evaluation of the data, mean, standard deviation, minimum and maximum values, frequency and percentage calculations, t-test and chi-square test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Speaks Turkish,
* 37-42 weeks gestation and in vaginal labor,
* The one with a single fetus and vertex development,
* Fetal weight between 2000-4000 gr,
* To have performed with mediolateral episiotomy,
* Pregnant women admitted to the delivery room,

Exclusion Criteria:

* Vacuum applied
* Forceps delivery
* Vaginal tear/ Disurge
* Anal sphincter damage
* Unusual need for lidocaine during episiotomy repair (more than 10ml)
* Intact perineum
* Any postnatal complications in the newborn.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
7 item perineal pain intensity measure | 3 hours
  Self-reported pain intensity before starting the first suturing, at the end of the 5th application, at the end of the 10th application, immediately after suturing was completed, and at 30 min, 60 min and 120 min after suturing was completed. Each item will be obtained using a visual analog scale. Each item is scored 0-10 (0=no pain; 10=unbearable pain).
Postpartum perineal pain intensity measure | 30 minutes
  Pain intensity will be determined 120 minutes after completion of stitching using the McGill scale form.There are 3 sections in the form. The first section consists of 15 descriptive words, 11 of which measure the sensory and 4 of which measure the perceptual dimension of pain. The words in the first section were rated on an intensity scale from 0 to 3 (0=None, 1=Mild, 2=Moderate, 3=Very). Three pain scores are obtained from this section: sensory pain score, perceptual pain score and total pain score. In the second section, the pain intensity of the person is measured with 5 word groups ranging from "mild pain" to "unbearable pain". In the third section, the current pain intensity of the patient is measured with a visual comparison scale.

SECONDARY OUTCOMES:
Postpartum comfort level | 30 minutes
  Based on the General Comfort Scale developed by Katharine Kolcaba in 1994, Karakaplan and Yıldız developed a postpartum comfort scale consisting of 34 items to determine postpartum comfort. This scale consists of three sub-dimensions: physical, psychospiritual and sociocultural. In order to evaluate the effect of acupressure application, only the physical sub-dimensions will be examined after two hours.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Deniz, PhD, Principal Investigator — TC Uskudar University; Ozlem Can Gurkan, Study Director — Marmara University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Solt Kirca A, Guducu N, Ikiz B. The Effect of Virtual Glasses Application on Pain and Anxiety During Episiotomy Repair: Randomized Controlled Trial. Pain Manag Nurs. 2023 Oct;24(5):e123-e130. doi: 10.1016/j.pmn.2023.06.004. Epub 2023 Jul 16. PMID 37455184
- [Result] Orhan M, Bulez A. The Effect of Virtual Reality Glasses Applied During the Episiotomy On Pain and Satisfaction: A Single Blind Randomized Controlled Study. J Pain Res. 2023 Jun 29;16:2227-2239. doi: 10.2147/JPR.S412883. eCollection 2023. PMID 37404226
- See also: The Effect of Virtual Glasses Application on Pain and Anxiety During Episiotomy Repair: Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/37455184/
- See also: The Effect of Virtual Reality Glasses Applied During the Episiotomy On Pain and Satisfaction: A Single Blind Randomized Controlled Study — https://pubmed.ncbi.nlm.nih.gov/37404226/